CLINICAL TRIAL: NCT00004090
Title: Gemcitabine (10 mg/m2/Min) and Cisplatin: A Phase I Study
Brief Title: Gemcitabine and Cisplatin in Treating Patients With Metastatic or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Albert B. Benson, MD, Northwestern University
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU CINJ98X1; NU-CINJ98X1; NCI-G99-1581
Record Dates: First submitted 1999-12-10; First posted 2004-08-30 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2011-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of gemcitabine and cisplatin in treating patients who have metastatic or recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of gemcitabine and cisplatin in patients with metastatic or recurrent nonhematologic malignancies.

OUTLINE: This is a dose escalation study of gemcitabine. Patients receive gemcitabine IV on days 1 and 8, followed immediately by cisplatin IV over 2 hours on day 8. Courses repeat every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-5 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 5 patients experience dose limiting toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 18 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic or recurrent nonhematologic malignancy that is not amenable to or has failed standard therapy Measurable or evaluable disease No uncontrolled brain metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: Neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Pulmonary: No respiratory failure Other: Not pregnant or nursing Fertile patients must use effective contraception No active infection or other concurrent severe medical illness that would interfere with compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas) and recovered No prior cisplatin or gemcitabine Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Cancer Institute of New Jersey, New Brunswick, New Jersey